CLINICAL TRIAL: NCT04616131
Title: Evaluating the Response to Neoadjuvant Chemotherapy With Circulating Tumor DNA in Pancreatic Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central DuPage Hospital (Other)
Collaborators: Elsa U. Pardee Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 21-012
Record Dates: First submitted 2020-10-21; First posted 2020-11-04 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-10

CONDITIONS: Pancreas Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
For patients who have been diagnosed with pancreatic cancer that has not spread outside of the pancreas and nearby lymph nodes. The purpose of this research study is to understand if we are able to detect pancreatic cancer DNA in the blood stream before, during, and after treatment.

DETAILED DESCRIPTION:
Cancer DNA in the blood stream is called circulating tumor DNA or ctDNA. The presence or absence of pancreatic cancer ctDNA in the blood stream may help clinicians to better understand pancreatic cancer behavior in response to specific treatments, like chemotherapy and surgery. Understanding how treatment alters the ctDNA can help future patients diagnosed with pancreatic cancer. The presence or absence of ctDNA or the clearance of ctDNA after treatment may help to guide further treatment decisions for cancer patients after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy or cytology proven adenocarcinoma of the pancreas
* No clinical evidence of metastatic disease on imaging
* Age 18 or older
* Receiving chemotherapy for non-metastatic pancreatic cancer

Exclusion Criteria:

* Biopsy proven metastatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female individuals age 18 and over planning to receive chemotherapy for pancreatic cancer that has not spread outside of the pancreas and nearby lymph nodes.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with circulating tumor DNA (ctDNA) levels as not detectable in their blood compared to number of patients with ctDNA detected. | 3 months
  Utilizing Tempus, a commercial laboratory ctDNA genetic profile panel investigators will analyze the number of patients who had detectable ctDNA in their blood prior to neoadjuvant chemotherapy who then had no detectable ctDNA after their chemotherapy treatment.

SECONDARY OUTCOMES:
Investigators will look for statistically significant correlations of ctDNA blood levels with clinical treatment responses of tumor grades, CA 19-9 units/milliliter blood level, and radiologic response by RECIST categories of complete response. | 12 months
  Association of ctDNA clearance with the following: pathologic treatment response per CAP tumor regression grade 0,1,2, and 3, blood level measurement of protein CA 19-9 units/milliliter, and radiologic response by tumor measurements in mm and using RECIST tumor measurement categories of complete response (CR), partial response (PR), stable disease (SD), and progressive disease (PD) for all patients, and margin assessment (R0/R1 resection) in resected patients.

CONTACTS AND LOCATIONS:
Overall Officials: Akhil Chawla, MD, Principal Investigator — Northwestern Medicine Central DuPage Hospital
Locations (3):
- United States (3):
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois

IPD SHARING:
Plan to Share IPD: No